CLINICAL TRIAL: NCT06435442
Title: A Phase 1 Study to Evaluate the Safety and PK/PD Drug-drug Interaction Between Epaminurad and Naproxen or to Assess the Safety and Multiple-Dose PK/PD Characteristics of Epaminurad in Healthy Volunteers
Brief Title: PK,PD and DDI of Epaminurad and Naproxen in Healthy Volunteers
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JW23103
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Healthy
MeSH Terms: interventions — Naproxen; URC102

STUDY DESIGN:
Intervention Model Description: PART 1: A open-label, multiple-dose, single group/ PART 2: A placebo-controlled, randomized, double-blind, multiple-dose, parallel group
Who Masked: Participant, Investigator
Masking Description: PART 1: None (Open Label)/ PART 2: Double (Participant, Investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): Epaminurad 6 mg, Epaminurad 9 mg, Naproxen 500 mg
  Interventions: Drug: Epaminurad, Naproxen
- Part 2(Test group) (Experimental): Epaminurad 6 mg, Epaminurad 9 mg
  Interventions: Drug: Epaminurad
- Part 2(Control group) (Placebo Comparator): Epaminurad 6 mg placebo, Epaminurad 9 mg placebo
  Interventions: Drug: Epaminurad placebo

INTERVENTIONS:
Drug: Epaminurad, Naproxen — Period 1: Epaminurad 6mg -> Epaminurad 9mg -> Epaminurad 9mg +Naproxen Period 2: Naproxen
  Other Names: URC102, Naxen
  Arms: Part 1
Drug: Epaminurad — Epaminurad
  Other Names: URC102
  Arms: Part 2(Test group)
Drug: Epaminurad placebo — Epaminurad placebo
  Other Names: URC102 placebo
  Arms: Part 2(Control group)

SUMMARY:
A Phase 1 Study to evaluate the safety, PK/PD, drug-drug interaction(DDI) of Epaminurad and Naproxen in Healthy Volunteers

DETAILED DESCRIPTION:
Part 1: to evaluate the safety, PK/PD, drug-drug interaction(DDI) of Epaminurad and Naproxen in Healthy Koreans/ Part 2: to evaluate the safety, PK/PD of Epaminurad in Healthy Caucasians

ELIGIBILITY:
Inclusion Criteria:

1. Age: 19~50
2. Weight: between 50.0 kg~90.0 kg, Body Mass Index(BMI): 18.0 kg/m^2 or heavier and below 30.0 kg/m^2
3. Part 1: Korean/ Part 2: Caucasian

Exclusion Criteria:

1. Medical history- chronic liver disease, acute gout attack, uric acid stone, diabetes, hypertension, hyperlipidemia or lipid abnormality
2. Clinical examination- eGFR (CKD-EPI) < 90mL/min/1.73m^2, Serum uric acid < 3 mg/dL or > 7 mg/dL, AST (SGOT), ALT (SGPT) > upper limit of normal ranges X 1.5, Total bilirubin, γ-GTP > upper limit of normal ranges X 1.5, CK > upper limit of normal ranges X 2, Positive serologic results Cystatin C > 1.26mg/L (man), > 1.19 mg/L (woman)

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 5 days
  To evaluate the AUC of Naproxen
Area under the plasma concentration versus time curve (AUC) | 7 days
  To evaluate the AUC of Epaminurad
Peak plasma concentrations (Cmax) | 7 days
  To evaluate the Cmax of Epaminurad
Peak plasma concentrations (Cmax) | 5 days
  To evaluate the Cmax of Naproxen

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-sang Yu, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No